CLINICAL TRIAL: NCT00225407
Title: A Double-Blind, Randomised, Placebo-Controlled, Cross-Over Study on the Pharmacokinetics and Effects of Cannabis
Brief Title: Processing and Effects of Cannabis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Collaborators: Netherlands: Ministry of Health, Welfare and Sports (Other Government)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: V/267002
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2005-09-23 (Estimated); Status verified 2005-03

CONDITIONS: Hypotension; Tachycardia
Keywords: Cannabis; Tetrahydrocannabinol; Pharmacokinetics; Psychomotor tests; Event related potentials
MeSH Terms: conditions — Hypotension; Tachycardia; Marijuana Abuse

INTERVENTIONS:
Drug: Smoking of cannabis cigarettes (different strength)

SUMMARY:
The purpose of this study is to investigate the processing of cannabis, and to investigate the occurrence of effects of cannabis on the cardiovascular system and the central nervous system; at higher levels of exposure.

DETAILED DESCRIPTION:
In Europe, cannabis is the most illicit used drug, mainly for its psychoactive properties (becoming "high" or "stoned"). The active compound in cannabis is THC (tetrahydrocannabinol). In recent years the strength of cannabis (marihuana) available on the market in the Netherland has increased (especially "netherweed"). The THC-content has increased from on average 8.6% in 2000 to on average 20.3% in 2004. Experienced users adapt their habit of smoking to the strength of the cannabis sigaret (joint). However, there is also a group of people, mainly young ones, who intent to smoke the joint entirely, and can therefore be exposed to higher levels of THC. Information is lacking about the effects of cannabis at higher levels of exposure. Because of this, the Ministry of Health, Welfare, and Sports of the Netherlands ordered the investigators to perform a study to gain more insight in this issue.

ELIGIBILITY:
Inclusion Criteria:

* Cannabis users (2-9 joints per month)

Exclusion Criteria:

* Psychiatric illness
* Evidence of excessive alcohol abuse
* Use of other drugs

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27
Dates: Start 2005-07; Study Completion 2005-12

PRIMARY OUTCOMES:
Serum concentration over time
Physical parameters (heart rate, blood pressure)
Psychomotor tests (such continuous attention)
Event related potentials

SECONDARY OUTCOMES:
Self-reporting questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Tjeert T Mensinga, MD, PhD, Principal Investigator — National Institute of Public Health and the Environment, the Netherlands
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

REFERENCES:
- [Derived] Hunault CC, Mensinga TT, Bocker KB, Schipper CM, Kruidenier M, Leenders ME, de Vries I, Meulenbelt J. Cognitive and psychomotor effects in males after smoking a combination of tobacco and cannabis containing up to 69 mg delta-9-tetrahydrocannabinol (THC). Psychopharmacology (Berl). 2009 May;204(1):85-94. doi: 10.1007/s00213-008-1440-0. Epub 2008 Dec 20. PMID 19099294